CLINICAL TRIAL: NCT04990024
Title: The Effect of Mediterranean or High Protein/Low Carbohydrate Diet on Arterial Stiffness in Non-diabetic, Obese Patients on Semaglutide: A Randomized Controlled Trial
Brief Title: The Effect of Different Diets on Arterial Stiffness in Obese Patients on Semaglutide
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Marlene Chakhtoura, Assistant Professor of Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2020-0136
Record Dates: First submitted 2021-07-02; First posted 2021-08-04 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: A computer-generated allocation sequence will be used, with a permuted block randomization (1:1). The biostatistician (MB) will generate the randomization sequence and will share it with a trial coordinator (MR) who is independent of the study team. Upon the recruitment of every participant, the study RA will contact the independent trial coordinator to receive the randomization code, in an opaque and sealed envelope.
  Randomization will take place at 1-30 days after starting Semaglutide. Treatment allocation will be in batches at the end of each month.
Masking Description: The design is open label as it is impossible to blind the participants and the research team for the study intervention. Each of the dietary interventions will be delivered in the format of intensive individual sessions about the diet, food selection and food recipes. Outcome assessors will be blind to the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Experimental): 30 participants will be randomized to this arm. The intervention consists of 8 visits, over a period of 24 weeks, including 6 individual educational sessions on Mediterranean diet in patients on Semaglutide and 2 reinforcement educational sessions towards the end of the trial. Dietary assessments and adherence questionnaires will be conducted on several visits to assess adherence.
  Interventions: Other: Dietary Intervention Med Diet
- High Protein/Low Carbohydrate Diet (Experimental): 30 participants will be randomized to this arm. The intervention consists of 8 visits, over a period of 24 weeks, including 6 individual educational sessions on High Protein/Low Carbohydrate diet in patients on Semaglutide and 2 reinforcement educational sessions towards the end of the trial. Dietary assessments and adherence questionnaires will be conducted on several visits to assess adherence.
  Interventions: Other: Dietary Intervention HP/LC Diet

INTERVENTIONS:
Other: Dietary Intervention Med Diet — The diet will consist of a calorie-restricted Med diet, with 500 Kcal/d energy restriction. The intervention consists of individual and reinforcement sessions on Med diet. During these sessions, the RA will go over the benefits of Med diet, what composition it should have, and how to make appropriate choices for meal planning, in addition to providing food lists, by season. The individual sessions with subjects will also allow to individualize the diet plan.
  Arms: Mediterranean Diet
Other: Dietary Intervention HP/LC Diet — This is a non-ketogenic diet consisting of ad libitum intake of proteins, fat, and vegetables, with restriction of daily carbohydrates to <130 g/d. The intervention consists of individual and reinforcement educational sessions on HP/LC, same as with Med diet (above). The individual sessions with subjects will also allow to individualize the diet plan.
  Arms: High Protein/Low Carbohydrate Diet

SUMMARY:
In patients initiating Semaglutide for weight management, the objective is to compare the effect of the Mediterranean diet and the high protein/low carbohydrate (HP/LC) diet CV parameters, namely arterial stiffness, measured by carotid-femoral pulse wave velocity (cfPWV), and visceral adipose tissue, in addition to other metabolic indicators.

DETAILED DESCRIPTION:
This is a 6-month open label pilot RCT that will be conducted on Lebanese subjects with obesity, upon the initiation of Semaglutide for medical weight management, as recommended by their physician. Patients will be randomized to 2 treatment arms: Med diet and HP/LC diet. Med diet will be hypocaloric, allowing the same energy restriction, of 500 Kcal/d, while the HP/LC diet will be ad libitum. Participants will be recruited from the Endocrine clinics at AUB-MC, and from satellite clinic next in Beirut. Brochures and posters of the trial will be available in the clinic waiting areas. Patients of both participating and non-participating physicians will be recruited in the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and premenopausal women, 18-49 years, with obesity defined as BMI ≥ 30 kg/m2
* Upon the initiation of Semaglutide (within the first 1-4 weeks) for medical weight management, for clinical purposes, as advised by the primary physician
* Able to commit for a 6-month trial visits

Exclusion Criteria:

* Pregnant women
* Patients who are taking or have taken other weight reducing drug therapies in the previous 6 months
* Patients who have undergone metabolic weight loss surgery
* Patients known to have diabetes (HbA1c ≥6.5% at screening)
* Patients with uncontrolled hypertension
* Patients with uncontrolled cardiac disease, pulmonary, renal or liver diseases, active cancer or psychiatric diseases
* Patients with excessive alcohol intake, defined as ≥ 2 glasses per day
* Patients known to have uncontrolled/ untreated thyroid disorders.
* Patients with cushing disease or polycystic ovaries, and those with neuro-endocrine or drug induced obesity (such as anti-psychotic, steroids, hormonal therapy): Such patients are resistant to weight loss, and they need treatment of their primary disease and/or cessation of the culprit medication to lose weight
* Patients with untreated gout
* Patients who have undergone bariatric surgery

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
cfPWV measurement and pulse wave analysis (PWA) using SphygmoCorCvMS V9 (AtCor Medical) | 6 months after enrollment
  Measured by an RA or a technician, based on the American Heart Association Council recommendations on arterial stiffness measurement in research. The distance from the suprasternal notch to the carotid pulse, and to the femoral site on the same side will be measured; the former distance is subtracted from the latter one. Ten seconds of carotid and 10 seconds of femoral arterial waveforms will be recorded, and the average of the data will be obtained for each of the sites.

SECONDARY OUTCOMES:
Body composition - visceral adipose tissue using dual x-ray absorptiometry (DXA) | 6 months after enrollment
  Measured by an RA or a technician, assessed using dual x-ray absorptiometry (DXA), Hologic machine, version 13.6.0.5, the preferred method for the assessment of body composition. The ISCD recommendations will be followed for body composition measurement.
Body composition - percent fat-free body mass using dual x-ray absorptiometry (DXA) | 6 months after enrollment
  Measured by an RA or a technician, assessed using dual x-ray absorptiometry (DXA), Hologic machine, version 13.6.0.5, the preferred method for the assessment of body composition. The ISCD recommendations will be followed for body composition measurement.
Body composition - percent body fat using dual x-ray absorptiometry (DXA) | 6 months after enrollment
  Measured by an RA or a technician, assessed using dual x-ray absorptiometry (DXA), Hologic machine, version 13.6.0.5, the preferred method for the assessment of body composition. The ISCD recommendations will be followed for body composition measurement.

OTHER OUTCOMES:
Dietary Assessment using 24-hour recalls | 6 months after enrollment
  Three-repeated 24-hour recalls (24 HR) administered via phone (2-week days and one week-end day, during one specific week). During the phone call, the participant will be asked to recall all what she/he has consumed during the past 24 hours, and the multiple pass approach of the USDA will be adopted.
Dietary Assessment using adherence questionnaires | 6 months after enrollment
  During the individual sessions, brief adherence assessment questionnaires for each diet, adapted from PREDIMED protocol, will be administered to calculate dietary adherence scores.
Anthropometric measurements - weight in kilograms, height in centimetres, aggregated into BMI (kilogram per meter squared). | 6 months after enrollment
  Weight and height will be measured following standard operating procedures (SOP) and BMI will be computed by dividing weight by height squared.
Anthropometric measurements - waist and hip circumference in centimetres, aggregated into waist to hip ratio ratio | 6 months after enrollment
  Waist and hip circumference will be measured following standard operating procedures (SOP).
Vital signs - blood pressure | 6 months after enrollment
  Blood pressure will be measured following standard operating procedures (SOP).
Vital signs - heart rate | 6 months after enrollment
  Heart rate will be measured following standard operating procedures (SOP).
Genetic studies | 6 months after enrollment
  Genetic studies will consist of Single Nucleoside Polymorphism (SNP) analysis of genes of the GLP1 receptors and cannabinoid receptor 1 will be performed in the molecular lab. These tests will be run at the endocrine core research Lab in batches at study completion.
Metabolic, inflammatory and appetite hormones in pg/mL | 6 months after enrollment
  Gastric inhibitory polypeptide (GIP), Leptin, Adiponectin, Orexin, IL6. These tests will be run at the endocrine core research Lab in batches at study completion.
Metabolic, inflammatory and appetite hormones in pmol/L | 6 months after enrollment
  Insulin and Ghrelin.These tests will be run at the endocrine core research Lab in batches at study completion.
Metabolic, inflammatory and appetite hormones in ng/mL | 6 months after enrollment
  Irisin and mineral hormones and markers, including Crosslaps, Osteocalcin, GLP1. These tests will be run at the endocrine core research Lab in batches at study completion.
Quality of Life Measurement as assessed by the SF-36 questionnaire | 6 months after enrollment
  SF-36 questionnaire filled by participant

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Chakhtoura, MD, MSc, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut - Medical Center, Beirut, Riad El Solh, Lebanon